CLINICAL TRIAL: NCT06123702
Title: Cannabidiol Effects on Fear Extinction in Social Phobia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HHC-2023-0022
Record Dates: First submitted 2023-11-02; First posted 2023-11-09 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Social Anxiety Disorder
Keywords: Cannabidiol, fear extinction
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to CBD or placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: Capsules will be in opaque bottles and the experimenter will not see the contents of the bottle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): 600 mg oral cannabidiol
  Interventions: Behavioral: Fear extinction; Drug: Cannabidiol Cap/Tab
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Behavioral: Fear extinction; Drug: Placebo

INTERVENTIONS:
Behavioral: Fear extinction — Extinction of conditioned fear response
Drug: Cannabidiol Cap/Tab — 12 50-mg capsules
  Other Names: CBD
  Arms: Cannabidiol
Drug: Placebo — 12 placebo capsules
  Arms: Placebo

SUMMARY:
The investigators will randomly assign participants with social anxiety disorder to receive oral cannabidiol (CBD) or placebo. Participants will undergo a fear conditioning and extinction trial, and the investigators will examine whether CBD increases the degree of fear reduction during extinction.

DETAILED DESCRIPTION:
This will be a double-blind, randomized controlled trial of cannabidiol (CBD) vs. placebo for potentiating fear extinction in adult outpatients with social anxiety disorder (SAD). After providing written informed consent and passing medical screening, participants will be assessed for SAD and other mental health concerns. They will then engage in a fear conditioning paradigm in which an electrical stimulation is applied to the wrist that is aversive but not painful (at a level determined by each participant) paired with pictures of angry faces. Following the fear conditioning paradigm, they will receive orally administered CBD or placebo. They will then undergo a fear extinction phase in which the conditioned angry faces are shown repeatedly with no further electrical stimulus. Fear toward the conditioned faces following extinction will be measured using galvanic skin response (GSR) and a visual analog scale of self-reported fear. The investigators predict that CBD, compared to placebo, will result in lower GSR and self-reported fear ratings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Any gender
3. Any race/ethnicity
4. Primary diagnosis of SAD according to the DIAMOND
5. At least moderate severity of SAD as evidenced by a DIAMOND severity rating of 4 (moderate) or higher
6. Able to speak, read and write English (this is necessary because the study measures are only validated in English)
7. Concurrent medications will be allowed so long as there is not a substantial risk of interaction with CBD
8. Able/willing to consent to participate in study

Exclusion Criteria:

1. <18 years old
2. Active substance use disorder or mania according to the DIAMOND
3. Severe risk of suicide or non-suicidal self-injury in the interviewer's judgment
4. Current or past schizophrenia spectrum disorder according to the DIAMOND
5. Developmental disability, including autism spectrum disorder, according to clinical interview
6. History of organic brain illness or head injury with loss of consciousness > 5 minutes
7. Liver function abnormalities as detected by liver functioning test
8. History of allergic reaction to CBD according to clinical interview
9. Unable or unwilling to abstain from CBD or tetrahydrocannabinol use for 24 hr prior to study participation
10. Pregnancy or lack of adequate contraception
11. Any clinical factors that would preclude the participant from providing informed consent or otherwise participating in the research, according to the interviewer's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin conductance | Single session (2.5 hours)
  Galvanic skin responses to conditioned stimuli
Distress ratings | Single session (2.5 hours)
  Subjective units of discomfort (0-100, 100 = maximum distress)

CONTACTS AND LOCATIONS:
Overall Officials: David Tolin, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Anxiety Disorders Center, Institute of Living, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No